CLINICAL TRIAL: NCT05827679
Title: Creation and Validation of a Clinical Evaluation Scale for Abdominal Condition of the Premature
Brief Title: Creation and Validation of a Clinical Evaluation Scale for Abdominal Condition of the Premature (ECAP)
Acronym: ECAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2022 COLNE; 2022-A02779-34 (Other: ANSM)
Record Dates: First submitted 2023-03-23; First posted 2023-04-25 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-04

CONDITIONS: Preterm Birth Complication; Digestive System Disease
Keywords: physiotherapy; abdominal massage
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Every year in France, 60,000 children are born prematurely (before 37 weeks of amenorrhea), and present an immaturity of their various systems, in particular the digestive system. This can result in feeding intolerance, which is expressed by abdominal distension, regurgitation or vomiting, irregular transit and abdominal discomfort. This feeding intolerance influences the length of hospitalization and can lead to necrotising enterocolitis, a major complication.

In the Neonatal Intensive Care Units of Clermont-Ferrand hospital center, abdominal massages have been performed by physiotherapists for several years in order to improve the condition of the digestive system. However, the indication for abdominal massage is very dependent on the caregivers in charge of the newborn and the evaluation of the abdominal condition remains subjective with a great variability between examiners. Thus, some newborns will receive massage multiple times a day while others will not.

Developmental care is essential for these premature infants, especially to avoid over-stimulation. It is important not to add care, such as massage, if it is not needed. It is therefore essential to properly assess the digestive status of premature babies in order to determine whether they have feeding intolerance and whether they require treatment with abdominal massage.

To date, the investigators have not found measurable criteria or existing scales that can describe the digestive status of newborns. The main objective of the study is therefore to create and validate a clinical assessment scale for the abdominal status of preterm infants.

DETAILED DESCRIPTION:
This is an observational study with longitudinal follow-up regarding the validation of a scale that the investigators have created.

Inclusions will be made when the patient arrives at the Clermont-Ferrand hospital center in the neonatal intensive care units. The patients will be evaluated daily from the 3rd day of life by the nurse, the physiotherapist and the resident of the service. The evaluation will be carried out at least 8 times over 21 days. If an abdominal massage is performed, an assessment of the abdominal condition by the scale will be necessary before and after each massage by the physiotherapist. Each assessment (by physio, nurse and resident) will be blinded and within a maximum time window of 30 minutes.

The first evaluator clears the patient's abdomen (clothing and diaper removed) and then performs the assessment of the abdomen blindly. A description has been written so that each evaluator can use the ECAP scale under the same conditions and with well-detailed judgment criteria in order to have an evaluation that is as reliable as possible.

The time taken to assess the premature baby's abdomen by the ECAP scale is less than 3 minutes. The evaluator fills out the ECAP assessment table, blindly.

Within the next 30 minutes (the patient's abdominal condition is considered stable during this time), the second and third assessors have to do the same.

These assessments are stored together with each patient's clinical data collection, and then analyzed by statisticians.

ELIGIBILITY:
Inclusion Criteria:

* newborns, born prematurely (before 37 weeks of amenorrhea)
* at least 3 days of life
* hospitalized in the neonatal intensive care units
* whose holders of parental authority are able to give free and informed consent to participate in this study

Exclusion Criteria:

* Newborns with congenital pathology such as malformation, genetic or chromosomal abnormality.
* Newborns whose holders of parental authority are protected by law (under guardianship) or under the age of 18.
* Rejection of participation by parents

Ages: 3 Days to 60 Days | Sex: All
Age Groups: Child
Study Population: Newborns born before 37 weeks of amenorrhea, hospitalized in the neonatal intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical Abdominal assessment scale for Preterm infant (ECAP scale) | up to 18 months
  score between 0 and 20

SECONDARY OUTCOMES:
Indication for abdominal massage on ECAP scale | up to 18 months
  score on the Clinical Abdominal assessment scale for Preterm infants, between 0 and 20 (higher scores meaning worse outcome)
ECAP scale validity | up to 18 months
  term of birth population
impact of massage on ECAP scale | up to 18 months
  variation of the score of Clinical Abdominal assessment scale for Preterm infants, between 0 and 20 (higher scores meaning worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Marie COLNÉ, Principal Investigator — mcolne@chu-clermontferrand.fr
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France